CLINICAL TRIAL: NCT04271124
Title: Comparison of Exercise Training
Brief Title: COPD and Inflammatory Mediators
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Acheche Amal, PhD, Faculty of Medicine, Sousse
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Effect of exercise training
Record Dates: First submitted 2020-01-30; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PR (Active Comparator)
  Interventions: Other: exercise training
- PR+ET (Experimental)
  Interventions: Other: exercise training

INTERVENTIONS:
Other: exercise training — The patients are allocated to PR+ET group or PR Each group receive an exercise training

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is widely spread all over the world. It is predicted to be the third leading cause of death by 2020.

DETAILED DESCRIPTION:
COPD is a common, preventable treatable disease that is characterized by an airflow limitation which is not fully reversible.Not only the long-term exposition to noxious particles and gases contributes to the development of COPD, but also many others factors such as genetics and cigarette smoking. Cigarettes are harmful and contribute to different extra pulmonary disorders. Although COPD affects lungs some extrapulmonary manifestations are prescribed such as muscle dysfunction, abnormal respiratory muscles and systemic inflammation. Indeed, the systemic inflammation[6, 8] is considered as a key process in the pathogenesis of COPD. It involves different cells and molecules; high levels of circulating of white blood cells, increased plasma c-reactive proteins (CRP), interleukin 6 (Il6) have been reported in.those patients.Likewise, systemic inflammation could worsen the comorbidities (cardiovascular, osteoporosis..) and may lead to the exercise limitation.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosed by pulmonary function testing
* Clinically stable
* Abscence of other obstructive diseases
* Signed written consent

Exclusion Criteria:

* Neuromuscular diseases -Severe psychiatric, neurologic or musculoskeletal conditions
* cardiovascular diseases.
* Contre-indications to physical therapy
* Acute exacerbations a month before the intervention

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change of Interleukins concentrations | Before the training, 2 months
  ELISA assay

SECONDARY OUTCOMES:
6Minutes Walk test | Before the training, 2 months
  patients performed the test

CONTACTS AND LOCATIONS:
Overall Officials: Yassine Trabelsi, professor, Study Director — Laboratoire de recherche:Physiologie de l'Exercice et Physiopathologie
Locations (1):
- Laboratoire de Recherche : Physiologie de l'Exercice et Physiopathologie, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No